CLINICAL TRIAL: NCT02908438
Title: Gonadotrophin Releasing Hormone Agonist Addition for Luteal Support in In-vitro Fertilization and Embryo Transfer Cycles
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-GnRHa for LPS
Record Dates: First submitted 2016-09-12; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: GnRHa;LPS

ARMS (2):
- GnRHa group (Experimental): Intervention: additional GnRHa for routine LPS GnRHa group receive three injections of GnRHa(Decapeptyl) ,0.1 mg s.c. on the day of ET, and D3 and D6 after ET in addition to routine LPS.
  Interventions: Drug: Gonadotrophin releasing hormone agonist(GnRHa)
- control group (No Intervention): Control group receive only the routine LPS.

INTERVENTIONS:
Drug: Gonadotrophin releasing hormone agonist(GnRHa) — GnRHa group receive three injections of GnRHa(Decapeptyl) ,0.1 mg s.c. on the day of ET, and D3 and D6 after ET in addition to routine LPS.
  Arms: GnRHa group

SUMMARY:
The study was designed to investigate the effect of luteal-phase administration of gonadotrophin releasing hormone agonist(GnRHa) on pregnancy outcomes in in-vitro fertilization-embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 37 years;
2. One or more high quality embryos have been got in IVF/ICSI treatment;
3. To transfer at lest 2 fresh embryos;
4. Uterine endometrial thickness ≥ 7mm;
5. Patients have signed informed consents.

Exclusion Criteria:

1. ≥3 IVF/ICSI/FET cycles and no pregnancy;
2. Polycystic ovary syndrome(PCOS);
3. uterine malformation;
4. endometriosis
5. patients with a history of recurrent pregnancy loss.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | up to 12 months